CLINICAL TRIAL: NCT03110458
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of 2 Dose Regimens of Orally Administered SENS-111 (100 mg and 200 mg) Given During 4 Days in Patients Suffering From Acute Unilateral Vestibulopathy
Brief Title: Efficacy of SENS-111 in Patients Suffering From Acute Unilateral Vestibulopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sensorion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SENS 111-201
Record Dates: First submitted 2017-03-27; First posted 2017-04-12 (Actual); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Acute Unilateral Vestibulopathy (AUV)
Keywords: Acute unilateral vestibulopathy, AUV
MeSH Terms: interventions — seliforant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SENS-111 100mg (Experimental): SENS-111 100mg: 2 Oral Dispersible Tablets (1 SENS-111 100 mg and 1 placebo)
  Interventions: Drug: SENS-111 100mg
- SENS-111 200mg (Experimental): SENS-111 200mg: 2 Oral Dispersible Tablets (SENS-111 100 mg)
  Interventions: Drug: SENS-111 200mg
- Placebo (Placebo Comparator): Placebo: 2 placebo Oral Dispersible Tablets
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: SENS-111 100mg — SENS-111 100mg is presented as 1 Oral Dispersible Tablet of SENS-111 100mg + 1 Oral Dispersible Tablet of placebo given twice on Day 1, second intake given approximately 12 hours (9 to 15 hours) after the first intake and thereafter given once daily on Days 2 to 5 inclusive. The corresponding total dose will be 500 mg for the entire study.
  Arms: SENS-111 100mg
Drug: SENS-111 200mg — SENS-111 200mg is presented as 2 Oral Dispersible Tablet of SENS-111 100mg given twice on Day 1,second intake given approximately 12 hours (9 to 15 hours) after the first intake and thereafter given once daily on Days 2 to 5 inclusive. The corresponding total dose will be 1000 mg for the entire study.
  Arms: SENS-111 200mg
Drug: Placebo Oral Tablet — Placebo is presented as 2 Oral Dispersible Tablets of placebo given twice on Day 1, second intake given approximately 12 hours (9 to 15 hours) after the first intake and thereafter given once daily on Days 2 to 5 inclusive. The corresponding total dose will be 0 mg for the entire study.
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of 2 dose-regimens of orally administered SENS-111 (100mg and 200mg) given during 4 days in patients suffering from Acute Unilateral Vestibulopathy (AUV)

ELIGIBILITY:
Inclusion criteria includes, but is not limited to:

* Subject has a diagnosis of definite Acute Unilateral Vestibulopathy

Exclusion criteria includes, but is not limited to:

* Acute continuous vertigo lasting more than 72 hours prior to randomization
* History of acute or chronic vestibular diseases
* History of prior acute central vestibular lesion
* Acute or chronic disease of middle ear

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael STRUPP, MD, Principal Investigator — University Hospital Munich
Locations (24):
- Columbia University Medical Center, New York, New York, United States
- University Hospital Hradec Králové, Hradec Králové, Czechia
- France (2):
  - CHU Gui de Chauliac, Montpellier
  - Hôpital Lariboisière, Paris
- Germany (4):
  - Kreiskliniken Altötting, Altötting, Bavaria
  - Klinikum Unfallkrankenhaus Berlin, Berlin
  - Universitätsklinikum Schleswig-Holstein Ratzeburger, Lübeck
  - Klinikum der Universität München, Munich
- Hungary (3):
  - Bajcsy-Zsilinszky Kórház és Rendelőintézet, Budapest
  - Pécsi Tudományegyetem, ÁOK Klinikai Központ, Pécs
  - Szegedi Tudományegyetem, Szent-Györgyi Albert Klinikai Központ, Szeged
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Care Campus, Haifa
  - Carmel Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
- Ospedale San Raffaele IRCCS, Milan, Italy
- South Korea (6):
  - Chonnam National University Hospital, Donggu
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Chungnam National University Hospital, Junggu
  - St. Paul's Hospital, The Catholic University of Korea, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo
Started | 37 | 36 | 34
Completed | 31 | 32 | 31
Not Completed | 6 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo | Total
Number analyzed (Participants) | 37 | 36 | 34 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (12.89) | 51.6 (14.14) | 51.1 (2.82) | 50.7 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 11 | 33
  Male | 23 | 28 | 23 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 21 | 19 | 60
  Unknown or Not Reported | 17 | 15 | 15 | 47
Body Weight [Mean (Standard Deviation); unit: Kg] | 82.2 (22.10) | 81.6 (18.9) | 80.1 (16.37) | 81.3 (18.94)

OUTCOME MEASURES:

1. Primary Outcome: Standing Vertigo Intensity
Description: The primary efficacy endpoint was the Area Under Curve (AUC) for the vertigo intensity measured by the Vertigo Intensity Visual Analogue Scale (VI-VAS) in standing position over the 4 treatment days (8 post-baseline assessments).
  The vertigo Intensity VAS is a non-anchored 10cm horizontal line. Patients were asked to rate the intensity of their vertigo making a vertical mark crossing the horizontal 10 cm line to indicate the severity from 0-100 when 0 indicates no severity and 100 indicates worse severity.
Time Frame: over the 4 treatment days
Population: Among the patients who started the study data was missing for some patients: 3 SENS-111 100mg, 1 SENS-111 200mg, 3 placebo patients
Measure: Mean (Standard Deviation); unit: mm*day
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo
Number analyzed (Participants) | 34 | 35 | 31
mm*day | 165.10 (71.02) | 155.10 (83.06) | 136.60 (62.61)
Statistical Analysis 1: Comparison: SENS-111 100mg vs SENS-111 200mg vs Placebo; Test type: Superiority; p = 0.8466, ANCOVA

2. Secondary Outcome: Worst Spontaneous Vertigo Intensity
Description: Worst spontaneous vertigo intensity measured by the AUC of the worst Vertigo Intensity Visual Analogue Scale (VI-VAS) over the 4 treatment days (8 post-baseline assessments).
  The vertigo Intensity VAS is a non-anchored 10cm horizontal line. Patients were asked to rate the intensity of their vertigo making a vertical mark crossing the horizontal 10 cm line to indicate the severity from 0-100 when 0 indicates no severity and 100 indicates worse severity
Time Frame: over the 4 treatment days
Population: Among the patients who started the study data was missing for some patients: 6 SENS-111 100mg, 4 SENS-111 200mg, 7 placebo
Measure: Mean (Standard Deviation); unit: mm*day
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo
Number analyzed (Participants) | 31 | 32 | 27
mm*day | 180.10 (67.20) | 170.40 (89.83) | 140.8 (64.66)
Statistical Analysis 1: Comparison: SENS-111 100mg vs SENS-111 200mg vs Placebo; Test type: Superiority; p = 0.9538, ANCOVA

3. Secondary Outcome: Proprioception D5
Description: The Romberg test assess the patient's ability to stand unassisted under 6 successive test conditions of increasing difficulty. In this test higher values are indicating a higher ability to stand unassisted, minimum total score is : 0 (impossibility to stand unassisted in any of the six conditions) and maximum is: 6. The change from Baseline of the total score of the six conditions of the Romberg test at the end of treatment (EOT) (Day 5) is evaluated.
Time Frame: End of treatment Day 5
Population: Among the patients who started the study data was missing for some patients: 5 SENS-111 100mg, 4 SENS-111 200mg, 8 placebo patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo
Number analyzed (Participants) | 32 | 32 | 26
score on a scale | 2.10 (1.46) | 2.00 (1.79) | 2.40 (1.45)
Statistical Analysis 1: Comparison: SENS-111 100mg vs SENS-111 200mg vs Placebo; Test type: Superiority; p = 0.3166, ANCOVA

4. Secondary Outcome: Proprioception D28
Description: The Romberg test assess the patient's ability to stand unassisted under 6 successive test conditions of increasing difficulty. In this test higher values are indicating a higher ability to stand unassisted, minimum total score is : 0 (impossibility to stand unassisted in any of the six conditions) and maximum is: 6. Change from Baseline of the total score of the six conditions of the Romberg test at the end of study (EOS) (Day 28) is evaluated.
Time Frame: End of study Day 28
Population: Among the patients who started the study data was missing for some patients: 7 SENS-111 100mg, 3 SENS-111 200mg, 8 placebo patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo
Number analyzed (Participants) | 30 | 33 | 26
score on a scale | 2.70 (1.60) | 3.00 (1.64) | 3.20 (1.46)
Statistical Analysis 1: Comparison: SENS-111 100mg vs SENS-111 200mg vs Placebo; Test type: Superiority; p = 0.393, ANCOVA

5. Secondary Outcome: Vestibular Spontaneous Nystagmus D5
Description: Change from Baseline of the Peak Slow Phase Velocity of the Peripheral Vestibular Spontaneous Nystagmus at the end of treatment (EOT) (Day 5). It is intended to record eye movements resulting from Nystagmus, measured by Oculography performed in complete darkness with visual fixation (10 seconds) or without fixation (30 seconds).
Time Frame: End of treatment Day 5 compared to basleine
Population: Among the patients who started the study data was missing for some patients: with fixation 13 SENS-111 100mg, 10 SENS-111 200mg, 11 placebo patients; without fixation 13 SENS-111 100mg, 13 SENS-111 200mg, 13 placebo patients
Measure: Mean (Standard Deviation); unit: degrees per second
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo
Number analyzed (Participants) | 24 | 26 | 23
degrees per second
  with fixation (10 seconds) | -2.30 (11.64) | -3.50 (10.27) | -5.7 (8.15)
  without fixation (30 seconds): number analyzed (Participants) | 24 | 23 | 21
  without fixation (30 seconds) | -1.2 (5.77) | -2.2 (7.22) | -2.7 (5.22)

6. Secondary Outcome: Vestibular Spontaneous Nystagmus D28
Description: Change from Baseline of the Peak Slow Phase Velocity of the Peripheral Vestibular Spontaneous Nystagmus at End of Study (Day 28). It is intended to record eye movements resulting from Nystagmus, measured by Oculography performed in complete darkness with visual fixation (10 seconds) or without fixation (30 seconds).
Time Frame: 28 days compared to baseline
Population: Among the patients who started the study data was missing for some patients: with fixation 11 SENS-111 100mg, 10 SENS-111 200mg, 12 placebo patients ; without fixation 12 SENS-111 100mg, 12 SENS-111 200mg, 13 placebo patients
Measure: Mean (Standard Deviation); unit: degrees per second
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo
Number analyzed (Participants) | 26 | 26 | 22
degrees per second
  with fixation (10 seconds) | -4.80 (15.10) | -7.9 (12.76) | -7.7 (11.59)
  without fixation (30 seconds): number analyzed (Participants) | 25 | 24 | 21
  without fixation (30 seconds) | -0.8 (8.84) | -2.9 (8.96) | -2.7 (6.50)

7. Secondary Outcome: Nausea Severity
Description: Nausea Severity measured by the Area under the Curve of the Nausea Intensity Visual Analogue Scale (NI-VAS).
  Patients were asked to rate the intensity of their nausea making a vertical mark crossing the horizontal 10 cm line to indicate the severity from 0-100 when 0 indicates no severity and 100 indicates worse severity.
Time Frame: over the 4 Treatment Days (Day 5)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm*day
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo
Number analyzed (Participants) | 34 | 35 | 31
mm*day | 93.00 (78.39) | 91.50 (79.73) | 92.60 (57.28)
Statistical Analysis 1: Comparison: SENS-111 100mg vs SENS-111 200mg vs Placebo; Test type: Superiority; p = 0.5324, ANCOVA

ADVERSE EVENTS:
Time Frame: up to end of study 28 days
Description: 104 subjects overall received any treatment and were included in the safety population (SENS-111 100 mg: 36 subjects,SENS-111 200 mg: 36 subjects and placebo: 32 subjects).
  Treatment emergent adverse events are displayed.
Arm/Group | SENS-111 100mg | SENS-111 200mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/36 | 0/32
Other Adverse Events (participants affected / at risk) | 4/36 | 5/36 | 7/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SENS-111 100mg (N=36) | SENS-111 200mg (N=36) | Placebo (N=32)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SENS-111 100mg (N=36) | SENS-111 200mg (N=36) | Placebo (N=32)
Extra dose administered (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (3) | 4 (6) | 7 (8)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT03110458/SAP_000.pdf
  • Study Protocol (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT03110458/Prot_001.pdf